CLINICAL TRIAL: NCT01903876
Title: Preventing Violence Against Women: A Web-based Approach
Brief Title: A Web-based Bystander Education Program
Acronym: RealConsent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura F Salazar, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00000472; R49CE000892 (NIH); EmoryVAW (Other: Other)
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Sexual Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Health promotion (Placebo Comparator): A 3-hour general mental health web-based program.
  Interventions: Behavioral: General Health Promotion
- Bystander & Sexual Violence Prevention (Experimental): A 3-hour web-based program designed to teach male college student bystanders to intervene.
  Interventions: Behavioral: Bystander & Sexual Violence Prevention

INTERVENTIONS:
Behavioral: Bystander & Sexual Violence Prevention — This 3-hour web-based program consists of six 30-minute modules that are interactive and range in number of segments (1-14) and types of activities. Each of the modules involves interactivity, didactic activities and two episodes of a serial drama, which allows for the modeling of positive behaviors and illustrate both positive and negative outcome expectations for intervening and for perpetrating abuse against women. Behaviors modeled include communicating with female sex partners, obtaining informed consent to have sex, and intervening to prevent abuse from taking place.
  Other Names: RealConsent
  Arms: Bystander & Sexual Violence Prevention
Behavioral: General Health Promotion — This general health promotion web-based program is 3-hours and provides a range of activities related to reducing day-to day stress and alleviating anxiety through meditation and exercise.
  Other Names: Stress & Mood Management
  Arms: General Health promotion

SUMMARY:
This is a study to determine whether a theoretically-driven web-based 3-hour intervention designed for male college students called RealConsent is effective in increasing prosocial intervening behaviors and in preventing sexual violence perpetration. Sexual violence programs for this population have been implemented for decades in the United States, but a program that is web-based and incorporates the bystander education model has never been implemented or tested. In this study, male college students will be recruited online, enrolled and randomly assigned to RealConsent or to a comparison condition. Prior to the intervention, investigators will ask questions about their intervening and sexually coercive behaviors and other theoretical and empirical factors related to the study outcomes. Investigators will survey the young men again at post-intervention, and at 6-months follow-up to determine whether young men in the RealConsent program intervened more often and engaged in less sexual violence compared to young men in the comparison condition. The main hypotheses are: (1) college men in the RealConsent program will report more instances of prosocial intervening; and (2) college men in the RealConsent program will report less sexual violence against women.

ELIGIBILITY:
Inclusion Criteria:

* Student matriculated at Georgia State University
* Male
* 18 to 24
* Undergraduate
* Self-identify as heterosexual or bisexual

Exclusion Criteria:

* Graduate student
* Self-identify as homosexual

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 743 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura F Salazar, PhD, Principal Investigator — Emory University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Salazar LF, Vivolo-Kantor A, Hardin J, Berkowitz A. A web-based sexual violence bystander intervention for male college students: randomized controlled trial. J Med Internet Res. 2014 Sep 5;16(9):e203. doi: 10.2196/jmir.3426. PMID 25198417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between Feb 2010 - April 2010.
Pre-assignment Details: N=368 participants completed the eligibility screener and provided informed consent in the study, but failed to complete the baseline assessment. Because our randomization occurred following completion of baseline assessment, these participants were not randomized to groups and were not included.
Period: Baseline to Post-Intervention Period
Arm/Group | General Health Promotion | Bystander & Sexual Violence Prevention
Started | 367 | 376
Completed | 183 | 268
Not Completed | 184 | 108
Not completed — Lost to Follow-up | 184 | 108
Period: Six-Month Follow-up Period
Arm/Group | General Health Promotion | Bystander & Sexual Violence Prevention
Started | 183 | 268
Completed | 92 | 123
Not Completed | 91 | 145
Not completed — Lost to Follow-up | 91 | 145

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Health Promotion | Bystander & Sexual Violence Prevention | Total
Number analyzed (Participants) | 367 | 376 | 743
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.33 (1.66) | 20.42 (1.69) | 20.38 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 367 | 376 | 743
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 12 | 23
  Asian | 73 | 73 | 146
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 83 | 83 | 166
  White | 200 | 208 | 408
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 367 | 376 | 743
Frequency of vaginal intercourse [Mean (Standard Deviation); unit: vaginal sex acts/60 days] | 8.38 (13.03) | 7.55 (12.75) | 7.96 (12.89)
Relationship status [Number; unit: participants] — Some data were missing for this variable; thus, the sum does not equal the overall numbers of baseline participants.
  participants
    Single | 270 | 289 | 559
    Married or has a partner | 6 | 1 | 7
    Engaged or committed | 87 | 82 | 169
    Separated | 0 | 0 | 0
    Divorced | 1 | 0 | 1
Legal knowledge of rape/assault [Mean (Standard Deviation); unit: units on a scale] — An index that assesses the level of knowledge regarding laws and policies on rape and sexual assault in Georgia and that ranges from 0 (no knowledge) to 9 (high levels of knowledge).
  units on a scale | 4.61 (1.78) | 4.54 (1.73) | 4.57 (1.75)
Knowledge of informed consent to have sex [Mean (Standard Deviation); unit: score on a scale] — This index measures the degree of knowledge regarding the elements of informed consent to have sex on a continuous scale with a range from 0 (no knowledge) to 14 (high level of knowledge).
  score on a scale | 11.46 (2.49) | 11.69 (2.44) | 11.58 (2.46)
Self-efficacy to intervene [Mean (Standard Deviation); unit: score on a scale] — This scale measures the degree of self-efficacy to intervene in situations that may contribute to a woman being sexually victimized. It is a continuous scale that ranges from 18 (no confidence) to 126 (high degree of confidence).
  score on a scale | 87.88 (23.6) | 88.74 (20.93) | 88.32 (22.27)
Intentions to intervene [Mean (Standard Deviation); unit: score on a scale] — This scale measures intentions to intervene in situations that place women at risk for sexual victimization. It is a continuous scale measure that ranges from 15 (no intentions to intervene) to 75 (high likelihood to intervene).
  score on a scale | 52.09 (12.78) | 52.68 (11.85) | 52.39 (12.3)
Outcome expectancies for intervening [Mean (Standard Deviation); unit: scores on a scale] — This scale measures the positive perceived outcomes that would likely occur if a participant intervened in a situation to prevent women from being sexually victimized. The scale is a continuous scale that ranges from 8 (low positive expectancies) to 40 (very positive expectancies).
  scores on a scale | 28.26 (4.86) | 28.72 (4.33) | 28.49 (4.6)
Self-comfort with men's inappropriate behaviors [Mean (Standard Deviation); unit: scores on a scale] — This scale measures men's level of comfort with other men's inappropriate behaviors toward women. The continuous scale ranges from 7 (not at all comfortable) to 49 (very comfortable).
  scores on a scale | 33.55 (10.71) | 32.68 (10.82) | 33.11 (10.76)
Rape myth acceptance [Mean (Standard Deviation); unit: scores on a scale] — The Illinois Rape Myth Acceptance Scale Short Form (IRMA-SF) was used to measure rape myths. This scale is a continuous scale measure with a range of 20 (no endorsement of rape myths) to 100 (high endorsement of rape myths).
  scores on a scale | 36.69 (10.29) | 35.88 (10.43) | 36.28 (10.36)
Outcome expectancies for engaging in rape [Mean (Standard Deviation); unit: scores on a scale] — This scale measures men's beliefs in positive outcomes for perpetrating sexual violence against a woman. The scale is continuous and ranges from 14 (no agreement with positive outcomes) to 70 (high degree of agreement with positive outcomes).
  scores on a scale | 58.02 (11.17) | 58.71 (10.76) | 58.37 (10.96)
Empathy for rape victims [Mean (Standard Deviation); unit: scores on a scale] — This scale is called the Rape Empathy scale and measures the degree of empathy for rape victims. The scale ranges from 19 (no empathy) to 95 (high level of empathy).
  scores on a scale | 68.78 (9.79) | 68.96 (9.66) | 68.87 (9.72)
Hostility towards women [Mean (Standard Deviation); unit: scales on a scale] — This is the Hostility Toward Women Scale that is a continuous measure that ranges from 0 (no hostility) to 10 (high degree of hostility).
  scales on a scale | 3.89 (2.54) | 3.42 (2.43) | 3.66 (2.49)
Date rape attitudes [Mean (Standard Deviation); unit: scores on a scale] — This is the Rape Attitudes and Beliefs Scale (RABS) that measures positive attitudes toward date rape. This continuous scale ranges from 50 (negative attitudes toward date rape) to 250 (very positive).
  scores on a scale | 128.45 (25.84) | 128.85 (24.07) | 128.65 (24.95)
Hyper-gender ideology [Mean (Standard Deviation); unit: scores on a scale] — Hypergender Ideology Scale Short Form (HGIS-S) is a continuous scale measure that assesses men's endorsement of masculine gender roles and ranges from 19 (no endorsement) to 95 (high degree of endorsement).
  scores on a scale | 46.38 (11.3) | 46.59 (11.28) | 46.49 (11.28)
Sexual coercion perpetration [Mean (Standard Deviation); unit: score on a scale] — This index is the Revised Conflict Tactics Scale (CTS-2): Sexual Coercion Subscale and assesses 7 sexually coercive-violent behaviors. The index ranges from 0 (no self report of sexually coercive behavior) to 7 (engaged in all of the behaviors).
  score on a scale | .76 (1.03) | .53 (1.07) | .64 (1.19)
Prosocial intervening [Mean (Standard Deviation); unit: percent scores on a scale] — This scale is the Reactions to Offensive Language and Behavior (ROLB) that measures whether or not men confronted inappropriate behaviors of other men. We used the 7-item self-behavior subscale plus an additional 8 items,which directly reflected the content of RealConsent. A series of 15 potential intervening situations were presented and participants were asked to indicate whether they had experienced the situation (yes/no), and whether they had intervened (yes/no). The scale ranges from 0% (did not intervene) to 100% (intervened each time).
  percent scores on a scale | 72 (24) | 72 (25) | 72 (24)

OUTCOME MEASURES:

1. Primary Outcome: Prosocial Intervening Behavior
Description: This scale is the Reactions to Offensive Language and Behavior (ROLB) index that measures whether or not men confronted inappropriate behaviors of other men. We used the 7-item self-behavior subscale plus an additional 8 items, which directly reflected the content of RealConsent. A series of 15 potential intervening situations were presented and participants were asked to indicate whether they had experienced this situation in past 6 months (yes/no), and whether they had intervened (yes/no). The scale ranged from 0% (did not intervene anytime) to 100% (intervened every time).
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percent score on a scale
Arm/Group | General Health Promotion | Bystander & Sexual Violence Prevention
Number analyzed (Participants) | 92 | 123
percent score on a scale | 72.2 (.031) | 81.1 (.028)
Statistical Analysis 1: Comparison: General Health Promotion vs Bystander & Sexual Violence Prevention; Test type: Non-Inferiority or Equivalence — equivalence; p = .044, ANCOVA

2. Secondary Outcome: Sexual Violence Perpetration
Description: This scale is the Conflict Tactics Scale revised, Sexual Coercion Subscale and assessed the number of sexually coercive/violent behaviors engaged in during the past 6 months. The index ranges from 0 (no engagement in any sexual violence) to 7 (engaged in all 7 sexually violent behaviors).
Time Frame: 6 months
Population: For some of the variables in this analysis, there were missing data. ANCOVA performed in SPSS will use a listwise deletion. This resulted in n=87 and n=115 for this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | General Health Promotion | Bystander & Sexual Violence Prevention
Number analyzed (Participants) | 87 | 115
score on a scale | .498 (.087) | .258 (.075)
Statistical Analysis 1: Comparison: General Health Promotion vs Bystander & Sexual Violence Prevention; Test type: Non-Inferiority or Equivalence — equivalence; p = .042, ANCOVA

ADVERSE EVENTS:
Arm/Group | General Health Promotion | Bystander & Sexual Violence Prevention
Serious Adverse Events (participants affected / at risk) | 0/367 | 0/376
Other Adverse Events (participants affected / at risk) | 0/367 | 0/376

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No